CLINICAL TRIAL: NCT06203054
Title: exClusion of the Left atrIal Appendage With PendITure™ (CLIP-IT) Post-Market Study
Brief Title: CLIP-IT Post-Market Study
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Medtronic Cardiac Surgery (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: MDT22049
Record Dates: First submitted 2024-01-02; First posted 2024-01-12 (Actual); Last update posted 2025-10-28 (Actual); Status verified 2025-10

CONDITIONS: Left Atrial Appendage Exclusion

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (1):
- Penditure™ Left Atrial Appendage (LAA) Exclusion System (Experimental): Penditure™ Left Atrial Appendage (LAA) Exclusion System
  Interventions: Device: Penditure™ Left Atrial Appendage (LAA) Exclusion System

INTERVENTIONS:
Device: Penditure™ Left Atrial Appendage (LAA) Exclusion System — Exclusion of the left atrial appendage using the Penditure™ Left Atrial Appendage (LAA) Exclusion System in subjects undergoing concomitant cardiac surgery.

SUMMARY:
The purpose of this study is to collect post-market clinical evidence on performance and clinical outcomes of the Penditure™ Left Atrial Appendage (LAA) Exclusion System in subjects undergoing concomitant cardiac surgery.

DETAILED DESCRIPTION:
Multi center, single-arm, nonrandomized, interventional, unblinded, post-market study. Up to 150 subjects will be enrolled and implanted with the Penditure™ Left Atrial Appendage (LAA) Exclusion Clip at up to 25 sites in the United States.

Subjects will be followed at 30 days, 3 months, 12-months and annually for 36-months.

ELIGIBILITY:
Inclusion Criteria:

* Patient is indicated to be treated with the Penditure™ left atrial appendage (LAA) Exclusion System
* Greater than or equal to 18 years of age
* The subject is willing and able to provide written informed consent and comply with study visit requirements

Exclusion Criteria:

* Prior left atrial appendage (LAA) isolation attempt(s)
* Need for emergent cardiac surgery
* Subject is contraindicated for multi-detector computed tomography (MDCT) and/or transesophageal echocardiogram (TEE)
* Life expectancy of less than 12 months
* History of cardiac surgery
* Pericarditis
* Presence of thrombus in the left atrium or left atrial appendage (LAA), prior to or during the procedure
* Patients requiring a heart transplant, insertion of a ventricular assist device or total artificial heart, and/or ascending aortic aneurysm or dissection repair requiring circulatory arrest
* Society of Thoracic Surgeons Predicted Risk of Mortality (STS-PROM) score greater than 4 or subject deemed to be high or extreme risk per surgeon assessment
* Ejection fraction less than 30%
* Chronic Kidney Disease Stage IV or V (estimated glomerular filtration rate (eGFR) <30 ml/min)
* New York Heart Association (NYHA) Class IV heart failure symptoms
* Patient has a documented history of substance (drug or alcohol) abuse
* Known allergy to device components (Nickel and/or Titanium)
* In the opinion of the investigator, the subject is not a suitable candidate for LAA isolation due to risks outweighing potential benefits including, complexity of planned concomitant procedures, or other pre-existing medical conditions
* Currently participating in an investigational drug or another device trial or study (excluding registries)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 150 (Actual)
Dates: Start 2024-02-26 (Actual); Primary Completion 2025-08-26 (Actual); Study Completion 2029-02 (Estimated)

PRIMARY OUTCOMES:
Rate of successful exclusion of the left atrial appendage (LAA) from the heart | 3 months post procedure
  The primary efficacy endpoint is the rate of successful exclusion of the left atrial appendage (LAA) from the heart defined as the absence of residual communication (≤ 3 mm residual contrast communication) between the left atrium (LA) and the left atrial appendage (LAA). For those successfully placed devices, exclusion will be confirmed at 3 months as demonstrated by multi-detector computed tomography (MDCT) scan.
Rate of device related adverse events | 30 days post procedure
  The primary safety endpoint is the composite rate of device-related serious adverse cardiac events at 30-days post-procedure.

SECONDARY OUTCOMES:
Rate of successful placement of the Penditure™ left atrial appendage (LAA) Exclusion System | At the time of procedure
  The secondary efficacy endpoint is defined as the rate of successful placement of the Penditure™ LAA Exclusion System defined as < 10 mm of residual stump proximal to the clip at the time of the procedure (measured by intraoperative TEE with doppler) without tissue damage requiring intervention.
Rate of device related adverse events | At 1 year, 2 year, and 3 years post procedure
  The secondary safety endpoint is defined as the composite device-related serious adverse cardiac event rate at 12-months and annually through 36 months.

CONTACTS AND LOCATIONS:
Locations (15):
- United States (15):
  - Emory Saint Joseph's Hospital, Atlanta, Georgia
  - Northwestern Memorial Hospital, Chicago, Illinois
  - Ascension St. Vincent Heart Center, Carmel, Indiana
  - University of Michigan Health System, Ann Arbor, Michigan
  - Corewell Health, Grand Rapids, Michigan
  - Mayo Clinic Saint Marys Campus, Rochester, Minnesota
  - Barnes Jewish Hospital, St Louis, Missouri
  - Saint Joseph's Hospital Health Center, Syracuse, New York
  - University Hospitals Cleveland Medical Center, Cleveland, Ohio
  - ProMedica Toledo Hospital, Toledo, Ohio
  - UPMC Pinnacle Harrisburg Campus, Harrisburg, Pennsylvania
  - University of Pittsburgh Medical Center UPMC Presbyterian, Pittsburgh, Pennsylvania
  - Lankenau Institute for Medical Research, Wynnewood, Pennsylvania
  - Houston Methodist Hospital, Houston, Texas
  - Swedish Medical Center Cherry Hill, Seattle, Washington